CLINICAL TRIAL: NCT03033771
Title: Evaluation of the Safety and Performance of the Multilayer Flow Modulator (MFM) for the Treatment of Chronic Type B Aortic Dissection
Brief Title: Dragon Study Europe
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiatis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-2015
Record Dates: First submitted 2017-01-19; First posted 2017-01-27 (Estimated); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Aortic Dissection Type B

STUDY DESIGN:
Intervention Model Description: Dragon Study Europe is an international, multicenter, prospective, non-randomized study. It is designed to evaluate safety and performance of the MFM for the treatment of chronic type B aortic dissection. About 35 patients in up to 11 countries will be enrolled and screened per the protocol-required inclusion, exclusion criteria, in order to obtain 30 completed patients. The main interim analysis, aiming at the early demonstration of safety and performance, will be performed after all patients included will complete their 6-month follow-up. A preliminary interim analysis will be performed on the first patients enrolled (15 completed patients) and with their 6-months follow-up available.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Patients presenting with chronic type B aortic dissection will have the MFM implanted.
  Interventions: Device: Implantation with the Multilayer Flow Modulator (MFM)

INTERVENTIONS:
Device: Implantation with the Multilayer Flow Modulator (MFM) — Endovascular implantation with the MFM
  Other Names: MFM, Multilayer Flow Modulator

SUMMARY:
Dragon Study Europe is an international, multicenter, prospective, non-randomized study. It is designed to evaluate safety and performance of the MFM for the treatment of chronic type B aortic dissection. About 35 patients in up to 11 countries will be enrolled and screened per the protocol-required inclusion, exclusion criteria, in order to obtain 30 completed patients. For early demonstration of safety and performance, an interim analysis report will be performed after all patients included will complete their 6-month follow-up.

The study purpose is to determine the safety and performance of the MFM for the endovascular treatment of chronic type B aortic dissection. It should be noted that the MFM has CE mark approval for aortic and peripheral artery aneurysms treatment.

DETAILED DESCRIPTION:
Aortic dissection (AD) is the surging of blood through a tear in the aortic intima with separation of the intima and media and creation of a false lumen.

The dissection may occur anywhere along the aorta and extend proximally or distally into other arteries. It occurs most commonly at the proximal ascending aorta (within 5 cm of the aortic valve) or the descending thoracic aorta (just beyond the origin of the left subclavian artery).

The passage of blood through the false channel can lead to complications such as spinal cord injury (paraplegia), lack of blood supply to the intestines (mesenteric ischemia) or lower extremities. The flow of blood in the false channel can cause these complications by pinching/narrowing off the flow of blood into the branches off the aorta. Aortic dissection always occurs in the setting of pre-existing degeneration of the aortic media. Causes include connective tissue disorders and injury. Atherosclerotic risk factors, notably hypertension, contribute in more than two thirds of patients.

Evidence of dissection is found in 1 to 3% of all autopsies. Population-based studies suggest that the incidence of AD is approximately 5-30 cases per million people per year. The diagnosis of AD is missed in 40% of cases on initial presentation, and 30% of AD are first diagnosed on post mortem exams.

African-Americans, men, the elderly, and people with hypertension are especially at risk. Peak incidence occurs at age 50 to 65 or, for patients with congenital connective tissue disorders (eg, Marfan syndrome, Ehlers-Danlos syndrome), at age 20 to 40.

Aortic dissections are classified anatomically, The DeBakey classification system is most widely used.

* Type I (50% of dissections): These dissections start in the ascending aorta and extend at least to the aortic arch and sometimes beyond.
* Type II (35%): These dissections start in and are confined to the ascending aorta.
* Type III (15%): These dissections start in the descending thoracic aorta just beyond the origin of the left subclavian artery and extend distally or, less commonly, proximally.

The Stanford system is simpler.

* Type A: These dissections involve the ascending aorta.
* Type B: These dissections are confined to the descending thoracic aorta. Patients with uncomplicated type B dissection have a 30-day mortality of 10%. Conversely, those who develop an ischemic leg, renal failure, visceral ischemia, or contained rupture often require urgent aortic repair; their mortality is 20% by day 2, and 25% by day 30.

For uncomplicated acute and chronic type B dissection, several series have shown that drug treatment alone can result in 78% three year survival after discharge from hospital. Current guidelines deem that the medical management remains the gold standard for uncomplicated type B aortic dissection and this benchmark is difficult to surpass. However, the medical treatment alone may put some patients at risk of serious complications such as progressive aortic enlargement, poor blood flow to some organs or the extremities, and aortic rupture.

The development of complicated dissection-defined by the presence of visceral or limb ischaemia, rupture, refractory pain, or uncontrollable hypertension-is the key factor that determines both intervention and outcome for patients with type B dissection.

Surgery is virtually always indicated if dissection involves the proximal aorta (type A dissection) and for complicated aortic dissection. In addition surgery may also be best for acute distal dissections in patients with Marfan syndrome. The goal of surgery is to obliterate entry into the false channel and reconstitute the aorta with a synthetic graft. Predictors of conventional surgery poor outcome include hypotension, renal failure, age > 70, abrupt onset of chest pain, pulse deficit, and ST-segment elevation on Electrocardiography.

TEVAR (Thoracic Endovascular Aortic Repair) aims to cover the primary entry tear in the descending aorta, resulting in a reduction of flow and pressure in the false lumen and formation of false lumen thrombosis.

Covered stent or bare stent reconstruction of branch vessels and re-entry tears, with false lumen thrombosis and remodelling. For acute (first 2 weeks) type B aortic dissection, the pooled early mortality rate was 6.4% with medical treatment and increased to 10.2% with TEVAR and 17.5% with open surgery, mostly for complicated cases. IRAD (International Registry of Acute Aortic Dissection) reported an in-hospital mortality rate of 32% for surgically treated individuals, 7% for those managed with endovascular techniques, and 10% for those managed with medical therapy alone. The in-hospital mortality rate of patients with complicated type B dissection was significantly higher after open surgery (33%) than after endovascular treatment (11%). This demonstrated that with appropriate use of endovascular stent graft placement, patients with complicated dissection enjoyed an improved prognosis, eventually similar to patients with an uncomplicated stable course requiring only medical management.

The presence of a rigid chronic dissection flap and multiple chronic re-entries often located distal to the treated thoracic aorta could have a negative impact on outcome. For patients with dissection extending into the abdominal aorta, TEVAR is seldom a definitive treatment, and the continued perfusion of the distal lumen could create further problems. The endovascular approach is associated with less morbidity and mortality. However, the longterm efficacy of an endovascular approach to preventing long-term aortic related death is still unclear.

Paraplegia and retrograde dissection are two of the most dreaded complications after TEVAR for type B dissection. Retrograde dissection occurs in 1% to 4% of patients and is more prevalent when the proximal landing zone is in the arch.

Spinal cord ischemia rates are lower after TEVAR than after open repair, but this complication remains a concern and has been reported in up to 4% of patients treated with TEVAR for chronic dissection. This result compare favourably with open repair, which has a reported 7% to 36% paraplegia risk.

Additionally, a significant proportion (12%-60%) of patients experience disease progression during follow-up after TEVAR, and thus requires further surgical procedures.

The Multilayer Flow Modulator® (MFM) (Cardiatis, Isnes, Belgium) has CE mark approval for peripheral/visceral and aortic aneurysms involving at least one branch. The aortic MFM is widely used for the thoracoabdominal aneurysm treatment. The clinical benefits of this technology have been suggested in studies about treatments of thoracoabdominal aneurysm, type B dissection, juxtarenal aortic aneurysm and peripheral artery aneurysm (celiac, hepatic, renal, iliac, subclavian). Also the prospective multicenter registry of peripheral and visceral aneurysms and the prospective multicenter STRATO Trial of TAAA, show good results at 12-month follow-up.

This MFM is an uncovered, self-expanding wire mesh with high radial force and flexibility. It is designed to modulate blood-flow dynamics by relieving local peak wall shear stress (PWSS), achieving stabilization of aneurysm-sac pressure and preserving side-branch patency.

In this study, the MFM® safety and performance will be evaluated in the use for the endovascular treatment of the chronic type B aortic dissection. Of course all patients were diagnosed according to standard of care and thoughtful decision before treatment/study intervention has to be made. In all cases the treating physician(s) shall consider and discuss alternative treatments with each individual patient before starting screening and enrolling into this study. Hence, once MFM® treatment within this study has been identified as feasible and desired mode of treatment with a state-of-the-art device with a beneficial risk benefit profile.

In general, treatment in this study will follow the routine course of an endovascular treatment of aortic pathologies, i.e. classical stenting procedures. Surgery, or stent-grafts are virtually always indicated if dissection involves the proximal aorta (type A dissection) and for complicated aortic dissection. In addition, surgery/stent-grafts may also be best for acute distal dissections in patients with congenital tissue disorders (non-exhaustively, such as Marfan, Loeys-Dietz or Ehler Danlos syndromes).

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Life expectancy > 12 months
* Informed consent understood, signed and patient agrees to all follow-up visits
* Chronic type B aortic dissection must be presenting with at least one of the following factors:

  * Uncontrollable hypertension
  * Persistent back/chest pain despite medical treatment
  * Expansion of aortic diameter (false lumen and total diameter)
  * With risk of progression, i.e. partial thrombosis of the false lumen
* Healthy proximal and distal landing zone
* Adequate arterial anatomy to perform EVAR by MFM
* Healthy branches and collaterals (no stenosis or previously treated by angioplasty)
* The patient must be available for the appropriate follow-up visits for the study duration

Exclusion Criteria:

* Stage 4 or 5 Renal Insufficiency as per K/DOQI clinical practice guidelines for chronic kidney disease (GFR < 29ml/min/1.73m²)
* Dissection or aneurysm rupture, impending or contained rupture
* Aortic root aneurysm
* Pleural effusion untreated at the procedure time
* Prior all surgical procedure within 30 days unless procedure is in preparation for device implantation or planned within 30 days post stent deployment
* Myocardial infarction or cerebral vascular accident within 6 weeks of treatment
* Presence/suspicion of connective tissue disorders, for example, Marfan or Ehlers-Danlos etc.
* Contraindications to the anticoagulant or/ and antiplatelet medications
* Thrombocytopenia
* Allergic reaction to a contrast agent
* Patient with undergoing or planned chemotherapy
* History of bleeding disorder (coagulopathy) or thrombophilia
* Patient with atrial fibrillation who are under anticoagulation therapy
* Presence/suspicion of infection (for example: mycotic aorta)
* The use of the MFM with stent-grafts or previously implanted stent-grafts
* Pregnant or breastfeeding woman
* Patients included in another clinical study
* Severe left ventricular dysfunction
* Significant arrhythmias
* Severe valvular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Re-establishment of the flow inside the true lumen | 30 days
  the re-establishment of the flow inside the true lumen will be evaluated using medical imagery. Data will be compaired to pre-op imaregy, and will be presented as a percentage of patient with true lumen repressurization compared to baseline.
Keeping all branches patent | 30 days
  the patency of branches emerging from the treated portion of the aorta will be evaluated and compared to pre-op data. Data will be presented as a percentage of branches patent per total number of branches involved in the diseased and treated portion of the aorta.
Re-establishment of the flow inside the true lumen | 12 months
  the re-establishment of the flow inside the true lumen will be evaluated using medical imagery. Data will be compared to pre-op imaregy, and will be presented as a percentage of patient with true lumen repressurization compared to baseline.
Keeping all branches patent | 12 months
  the re-establishment of the flow inside the true lumen will be evaluated using medical imagery. Data will be compaired to pre-op imaregy, and will be presented as a percentage of patient with true lumen repressurization compared to baseline.

SECONDARY OUTCOMES:
Mortality at 30 days | 30 days
  Percentage of patients deceased at 30 days
Number of Serious Adverse Events | 30 days, 12 months, 24 months and 36 months
Technical Success | The technical success is evaluated/recorded post-procedure and presented in the 12 months report
  Successful delivery and deployment of the MFM
Procedural/in-hospital evaluations (Anesthesia time) | The Procedural/in-hospital evaluation are recorded during hospital stay and collected data is presented in the 12 months report.
  descriptive statistics on Anesthesia time (min)
Procedural/in-hospital evaluations (Fluoroscopy time) | The Procedural/in-hospital evaluation are recorded during hospital stay and collected data is presented in the 12 months report.
  Descriptive Statistics on fluoroscopy time (min)procedure time; time to hospital discharge
Procedural/in-hospital evaluations (Contrast Volume) | The Procedural/in-hospital evaluation are recorded during hospital stay and collected data is presented in the 12 months report
  Descriptive Statistics on contrast volume (ml)
Procedural/in-hospital evaluations (Estimated Blood loss) | The Procedural/in-hospital evaluation are recorded during hospital stay and collected data is presented in the 12 months report.
  Descriptive Statistics on contrast Estimated Blood loss (ml)
Procedural/in-hospital evaluations (procedure time) | The Procedural/in-hospital evaluation are recorded during hospital stay and collected data is presented in the 12 months report.
  Descriptive Statistics on procedure time (min)
Procedural/in-hospital evaluations (time to hospital discharge) | The Procedural/in-hospital evaluation are recorded during hospital stay and collected data is presented in the 12 months report.
  Descriptive Statistics on time to hospital discharge (days).

CONTACTS AND LOCATIONS:
Overall Officials: Victor Costache, MD PhD, Principal Investigator — Sanador Hospital, Bucharest, Romania
Locations (4):
- Bulgaria (2):
  - City Clinic Burgas, Burgas
  - City Clinic Sofia, Sofia
- Romania (2):
  - Sanador Hospital, Bucharest
  - European Hospital Polisano, Sibiu

IPD SHARING:
Plan to Share IPD: No